CLINICAL TRIAL: NCT00220467
Title: Cognitive Effects of Aerobic Exercise for Adults With Mild Cognitive Impairment: A Controlled Trial
Brief Title: Cognitive Effects of Aerobic Exercise for MCI Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: Alzheimer's Association (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDIS 0008; ALZ ASSOC BL18 (SIBCR)
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Mild Cognitive Impairment
Keywords: MCI; aging; cognition; exercise; aerobic; insulin
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Aerobic exercise

SUMMARY:
The specific aims for the study will be to determine if aerobic exercise enhances cognition for older adults who are at greater risk for developing Alzheimer's disease, and to evaluate whether change in insulin sensitivity predicts cognitive performance for subjects randomized to the aerobic exercise group. Sedentary older adults diagnosed with mild cognitive impairment will participate in a 6-month supervised protocol of either aerobic exercise or stretching. Cognitive testing and blood collection will occur at baseline, and months 3 and 6. Before and after the 6-month intervention, insulin sensitivity, maximum aerobic capacity, and body fat composition and distribution (via CT scan) will be assessed for all subjects. The results of this study may provide support for a relatively simple and inexpensive treatment strategy that specifically targets many of the health factors that directly influence risk of cognitive decline for older adults.

DETAILED DESCRIPTION:
The specific aims for the study are 1) to determine if aerobic exercise enhances cognition for older adults with mild cognitive impairment, 2) to evaluate whether change in insulin sensitivity predicts cognitive performance for subjects in the aerobic exercise group, and 3) to relate exercise effects on insulin sensitivity and cognition to growth factor expression, inflammatory markers, catecholamines, beta-amyloid, and body-fat composition. Using a randomized controlled parallel group design, 40 sedentary older adults diagnosed with mild cognitive impairment will participate in a 6-month supervised protocol of either aerobic exercise or stretching. Cognitive testing and blood collection will occur at baseline, and months 3 and 6. Before and after the 6-month intervention, insulin sensitivity (via hyperinsulinemic-euglycemic clamp), maximum aerobic capacity (via respiratory gas exchange and cardiopulmonary fitness measures), and body fat composition (via DEXA scan) and distribution (via CT scan) will be assessed for all subjects. The results of this study may provide support for a relatively simple and inexpensive treatment strategy that specifically targets many of the health factors that directly influence risk of cognitive decline for older adults.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with mild cognitive impairment, at least 55 years of age, sedentary (elevated HR & SOB <3x/wk and <30min on each occasion), overall good general health, willing to exercise at least 4 times/wk for 6 months

Exclusion Criteria:

* Significant neurologic disease that might affect cognition, such as a diagnosis of Alzheimer's disease, stroke, Parkinson's disease, multiple sclerosis, or severe head injury with loss of consciousness; significant medical illness or organ failure such as liver disease, significant elevations in liver function tests, kidney disease, uncontrolled hypertension (BP>140/90 on medication); cardiovascular disease defined as any acute cardiovascular abnormality, such as new or unstable angina, uncontrolled irregular heart beat (treated a-fib and occasional PVC's are OK) or symptomatic heart failure, acute shortness of breath for any reason, or clinically significant edema; chronic lung disease, or musculoskeletal impairment (impaired walking); current use of anti-psychotic, anti-convulsant, anti-coagulant, sedative, or any cognition-enhancing medications; current or previous use of hypoglycemic agents or insulin.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-01; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change in cognitive scores
Change in insulin sensitivity

SECONDARY OUTCOMES:
Change in biomarkers associated with Alzheimer's disease progression
Correlation between cognitive scores, insulin sensitivity, & biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Baker, PhD, Principal Investigator — VA Puget Sound Health Care System; University of Washington
Locations (2):
- United States (2):
  - Veterans Affairs Puget Sound Health Care System, Seattle, Washington
  - Veterans Affairs Puget Sound Health Care System, Tacoma, Washington